CLINICAL TRIAL: NCT00000930
Title: Infected Participants Protocol: Evaluation of Natural History of HIV Infection in Newly HIV-Infected Persons in HIVNET Target Populations
Brief Title: A Study of HIV in Newly Infected Individuals
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: HIVNET 019
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Sexual Partners; Drug Resistance, Microbial; Cohort Studies; Risk Factors; Substance Abuse, Intravenous; Disease Progression; Homosexuality, Male; Genotype; Phenotype
MeSH Terms: conditions — HIV Infections; Substance Abuse, Intravenous; Disease Progression; Homosexuality, Male

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens appropriate for clinical and laboratory assessments and necessary for evaluation of study outcome measures

GROUPS / COHORTS (2):
- A: HIV-infected individuals enrolled in HIVNET D01
- B: Individuals with newly acquired HIV infection

SUMMARY:
The purpose of this study is to see how HIV reacts in the immune systems of patients who have recently been infected with HIV. This study also examines HIV's resistance to anti-HIV drugs in newly infected patients.

Certain populations are good candidates for participation in HIV vaccine trials. These groups include men who have sex with men, IV drug users, and women at risk of getting HIV through heterosexual contact. Learning how HIV behaves in these populations once they become infected can help with the planning of future HIV vaccine studies.

DETAILED DESCRIPTION:
This study provides an opportunity to prospectively monitor markers of HIV infection and disease progression in cohorts suitable for HIV vaccine trials. The detection of changes in HIV phenotype and genotype, clinical progression rates, and antiretroviral resistance within study populations over time are important for planning future HIV vaccine trials.

This study consists of two parts. Part A includes HIV-infected patients who enrolled in HIVNET D01.1 (infected-participants cohort of HIVNET D01) and whose HIV disease has been closely monitored and characterized. This study continues to monitor these patients with follow-up evaluations every 3 months for the first 18 months and then every 6 months thereafter. Part B includes newly HIV-infected patients. These patients are monitored with clinical and laboratory evaluations at 0, 1, 3, 6, 9, 12, and 18 months, and then every 6 months through Year 5.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection, as documented by enrollment in HIVNET D01.1 (Part A patients) or by standard HIV serological tests or demonstrated HIV infection on virologic assay (Part B patients).

Part A only:

* Previous enrollment in infected-participants cohort of HIVNET D01.

Part B only:

* Initial HIV-seronegativity on an HIVNET protocol (other than an HIV vaccine protocol) and testing positive for HIV at a subsequent clinic visit.
* Confirmation of HIV infection and documentation of HIV negative antibody test within 8 months of first positive test.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* An obvious psychological/psychiatric disorder that would invalidate the informed consent process or otherwise contraindicate participation in the study.

Prior Medication:

Excluded:

* Participation in a HIVNET HIV vaccine trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Dates: Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Detection of changes in HIV phenotype and genotype | Throughout study
Clinical progression rates | Throughout study
Antiviral resistance | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Celum C, Study Chair; Buchbinder S, Study Chair; Sheppard H, Study Chair
Locations (12):
- United States (12):
  - Los Angeles County / Health Research Assoc / Drew Med Ctr, Los Angeles, California
  - San Francisco Dept of Hlth / AIDS Office, San Francisco, California
  - Denver Dept of Public Health / HIVNET, Denver, Colorado
  - Univ of Illinois Chicago / Howard Brown Hlth Ctr, Chicago, Illinois
  - Johns Hopkins Univ, Baltimore, Maryland
  - Fenway Community Health Ctr / HIVNET, Boston, Massachusetts
  - New York Univ Med Ctr, New York, New York
  - Bronx-Lebanon Hosp Ctr, The Bronx, New York
  - New York Blood Ctr, The Bronx, New York
  - Univ of Pennsylvania / HIVNET, Philadelphia, Pennsylvania
  - Miriam Hosp, Providence, Rhode Island
  - Univ of Washington, Seattle, Washington